CLINICAL TRIAL: NCT01177215
Title: Implementation of an Adaptive Algorithm to Improve Chest Tube Therapy in Patients With Pulmonary Leaks Following Thoracic Surgery
Brief Title: Investigation of an Adaptive Treatment Algorithm for Post-op Thoracic Patients to Reduce the Length of Drainage
Acronym: AATD
Status: Terminated | Type: Observational
Why Stopped: Interim analysis showed that the tested protocol did not improve treatment
Sponsor: Medela AG (Industry)
Responsible Party: Principal Investigator, Inez Cregan, Study Director, Medela AG
Other Study IDs: GE-ADAPTALGO-2010
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Fistula
Keywords: Algorithm; Treatment Protocol; Thoracic Drainage Device
MeSH Terms: interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Digital chest tube: All patients will be treated with the digital chest tube device
  Interventions: Procedure: Thoracic Surgery

INTERVENTIONS:
Procedure: Thoracic Surgery — Wedge Resection Segmental Resection Lobectomy
  Other Names: Thopaz Drainage Device

SUMMARY:
The purpose of this study is to reduce the length of drainage using a treatment protocol to control the manipulation of the applied vacuum to the pleural cavity.

DETAILED DESCRIPTION:
In this prospective study, a treatment algorithm is tested in a subgroup of patients with postoperative pulmo-pleural fistula. The primary aim is to reduce the duration of pulmo-pleural fistulation. Secondary aim is to reduce the duration of chest tube therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a post operative air leak after 16 to 24 hours bigger than 50ml/min.

Exclusion Criteria:

* Patients with an empyema
* Patients with a spontaneous pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic Surgery Patient
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Duration of pulmo-pleural fistulation | July 2011 - March 2012
  The duration of a postoperative pulmo-pleural fistula is monitored.

SECONDARY OUTCOMES:
Duration of Chest tube therapy | July 2011 - March 2012
  Duration of postoperative chest tube therapy is monitored.
Applicability of a diagnostic "Leakage Scale" | July 2011 - March 2012
  Applicability of a generated scale that categorizes the pulmonary air leak is tested.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Walles, MD FETCS, Principal Investigator — Schillerhoehe Hospital
Locations (4):
- Germany (4):
  - Klinikum Bremen-Ost, Bremen, City state Bremen
  - Klinik Schillerhöhe, Gerlingen, Gerlingen
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Krankenhaus Großhansdorf, Großhansdorf

REFERENCES:
- [Background] Alex J, Ansari J, Bahalkar P, Agarwala S, Rehman MU, Saleh A, Cowen ME. Comparison of the immediate postoperative outcome of using the conventional two drains versus a single drain after lobectomy. Ann Thorac Surg. 2003 Oct;76(4):1046-9. doi: 10.1016/s0003-4975(03)00884-1. PMID 14529982
- [Background] Baumann MH. What size chest tube? What drainage system is ideal? And other chest tube management questions. Curr Opin Pulm Med. 2003 Jul;9(4):276-81. doi: 10.1097/00063198-200307000-00006. PMID 12806240
- [Background] Brunelli A, Sabbatini A, Xiume' F, Refai MA, Salati M, Marasco R. Alternate suction reduces prolonged air leak after pulmonary lobectomy: a randomized comparison versus water seal. Ann Thorac Surg. 2005 Sep;80(3):1052-5. doi: 10.1016/j.athoracsur.2005.03.073. PMID 16122484
- [Background] Cerfolio RJ, Bryant AS. The benefits of continuous and digital air leak assessment after elective pulmonary resection: a prospective study. Ann Thorac Surg. 2008 Aug;86(2):396-401. doi: 10.1016/j.athoracsur.2008.04.016. PMID 18640304
- [Background] Varela G, Jimenez MF, Novoa NM, Aranda JL. Postoperative chest tube management: measuring air leak using an electronic device decreases variability in the clinical practice. Eur J Cardiothorac Surg. 2009 Jan;35(1):28-31. doi: 10.1016/j.ejcts.2008.09.005. Epub 2008 Oct 9. PMID 18848460